CLINICAL TRIAL: NCT00422721
Title: Genetical, Multi-center, Prospective Study of Phenotyping and Genotyping of Patients Suffering From Congenital Amaurosis of Leber or From an Early Severe Retinal Dystrophy in the Aim of the Realisation of a Clinical Trial of Gene Therapy
Brief Title: Genetic Study of Patients Suffering From Congenital Amaurosis of Leber or From an Early Severe Retinal Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD 06/8-F; ID RCB 2006-A00192-49
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Amaurosis; Retinal Diseases
Keywords: early severe retinal dystrophy; amaurosis of leber
MeSH Terms: conditions — Blindness; Retinal Diseases; Retinal Dystrophies | interventions — Refractometry; Wechsler Scales; Visual Fields; Color Vision; Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: realization of a family tree
Procedure: refractometry
Procedure: evaluation of the presence of a nystagmus
Procedure: ocular behavior
Procedure: test of baby vision
Procedure: test of keenness
Procedure: reading test
Procedure: visual field
Procedure: color vision
Procedure: electroretinographical activity
Procedure: biomicroscopical test
Procedure: retinal imaging
Procedure: retinal autofluorescence
Procedure: genotyping

SUMMARY:
Retinal dystrophies are responsible for numerous cases of blindness, and there are no therapeutic possibilities today. Gene therapy is efficient in a dog model concerning dystrophy linked to a mutation of the rpe65 gene. If such a therapy is to be considered for humans, it is urgent to select, at a national level, patients suffering from dystrophy linked to a mutation of the rpe65 gene. The systematic correlation of phenotype/genotype is an anatomical-functional approach, but it also identifies patients who may be potentially included in a future gene therapy study. Indeed, identification of people with a mutation of rpe65 is still insufficient in France (compared to other European countries) because of a lack of systemic genotyping of retinal dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical characteristics of amaurosis of Leber
* Patients suffering from an early severe retinal dystrophy
* Patients with social insurance
* Patients with a consent form signed

Exclusion Criteria:

* Retinal dystrophy with autosomal dominant transmission
* Retinal dystrophy occuring after 5 years of age
* Syndromical retinal dystrophy with one or more systemic manifestations
* Familial macular degeneration
* Familial choroid dystrophy
* Non-degenerative retinopathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Michel Weber, MD, Principal Investigator — Nantes University Hospital; Sabine Defoort, MD, Principal Investigator — CHU de Lille; Bernard Puech, MD, Principal Investigator — CHU de Lille; Isabelle Drumaré, MD, Principal Investigator — CHU de Lille; Christian Hamel, MD, Principal Investigator — CHU de Montpellier; Carl Arndt, MD, Principal Investigator — CHU de Montpellier; Olivier Roche, MD, Principal Investigator — Hôpital Necker; Christophe Orssaud, MD, Principal Investigator — Hôpital Necker; Emmanuel Bui Quoc, MD, Principal Investigator — Hôpital Necker; Saddek Mohand Saïd, MD, Principal Investigator — CNO XV-XX; José-Alain Sael, MD, Principal Investigator — CNO XV-XX; Hélène Dollfus-Waltmann, MD, Principal Investigator — CHU de Strasbourg
Locations (1):
- CHU de Nantes, Nantes, France